CLINICAL TRIAL: NCT01129271
Title: A Randomized, Placebo-controlled, Two-sequence, Two-period Crossover Study, to Investigate a Potential Food Effect on the Pharmacodynamic and Bioavailability of Repeated Oral Doses of Clopidogrel (300 mg Loading Dose Followed by 75 mg/Day) in Healthy Male Subjects
Brief Title: Food Effect Study on Pharmacodynamic and Bioavailability of Clopidogrel 300/75 mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ALI11209
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group clopidogrel fed - fasting (Experimental): Period 1:
  * Day 1: clopidogrel 300 mg loading dose with high fat breakfast
  * Day 2 to Day 5: clopidogrel 75 mg/day with standard breakfast, once daily
  Period 2:
  * Day 1: clopidogrel 300 mg loading dose under fasted conditions
  * Day 2 to Day 5: clopidogrel 75 mg/day under fasted conditions, once daily
  Interventions: Drug: clopidogrel
- Group placebo fed - fasting (Placebo Comparator): Period 1:
  * Day 1: placebo loading dose with high fat breakfast
  * Day 2 to Day 5: placebo with standard breakfast, once daily
  Period 2:
  * Day 1: placebo loading dose under fasted conditions
  * Day 2 to Day 5: placebo under fasted conditions, once daily
  Interventions: Drug: Matching placebo
- Group clopidogrel fasting - fed (Experimental): Period 1:
  * Day 1: clopidogrel 300 mg loading dose under fasted conditions
  * Day 2 to Day 5: clopidogrel 75 mg/day under fasted conditions, once daily
  Period 2:
  * Day 1: clopidogrel 300 mg loading dose with high fat breakfast
  * Day 2 to Day 5: clopidogrel 75 mg/day with standard breakfast, once daily
  Interventions: Drug: clopidogrel
- group placebo fasting -fed (Placebo Comparator): Period 1:
  * Day 1: placebo loading dose under fasted conditions
  * Day 2 to Day 5: placebo in fasted conditions, once daily
  Period 2:
  * Day 1: placebo loading dose with high fat breakfast
  * Day 2 to Day 5: placebo with standard breakfast, once daily
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: clopidogrel — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Group clopidogrel fasting - fed; Group clopidogrel fed - fasting
Drug: Matching placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Group placebo fed - fasting; group placebo fasting -fed

SUMMARY:
Primary objective:

* Investigate the potential food effect on Adenosine diphosphate(ADP)-induced platelet aggregation after 5-day repeated doses of clopidogrel (300 mg loading dose followed by 4 days 75 mg/day) in healthy subjects

Secondary objectives are to investigate the potential food effect on:

* ADP-induced platelet aggregation after 300 mg loading dose of clopidogrel
* Pharmacokinetic profiles of clopidogrel and its active metabolite after 5-day repeated doses of clopidogrel

DETAILED DESCRIPTION:
The total duration per subject is 8-9 weeks broken down as follows:

* Screening: 2 to 21 days before the first dosing
* Fed period: 7 days including 5 treatment days
* Washout: at least 14 days after last dosing
* Fasted period: 7 days including 5 treatment days
* End of study: 7 to 10 days after the last dosing

ELIGIBILITY:
Inclusion Criteria:

Healthy male subjects:

* as determined by medical history, physical examination including vital signs and clinical laboratory tests
* with a body weight between 50kg and 95 kg and a Body Mass Index (BMI) between 18 and 30 kg/m2

Exclusion Criteria:

* Evidence of inherited disorder of coagulation/hemostasis functions
* Smoking more than 5 cigarettes or equivalent per day
* Abnormal hemostasis screen
* Any contraindication to clopidogrel
* Unability to abstain from intake of any drug affecting haemostasis throughout the whole study duration

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum platelet aggregation intensity (MAI) induced by Adenosine diphosphate (ADP) 5µM after 5 days treatment | Day 5 of each period

SECONDARY OUTCOMES:
Maximum platelet aggregation intensity (MAI) induced by ADP 5µM after loading dose and high fat breakfast | 6 hours and 24 hours after first dosing of each period
Clopidogrel pharmacokinetic parameters (maximum plasma concentration (Cmax) and area under the plasma concentration curve (AUC0-24)) after 5 days treatment | up to 24 hours postdose on Day 5 for each period
Clopidogrel active metabolite pharmacokinetic parameters (Cmax and AUC0-24) after 5 days treatment | up to 24 hours postdose on Day 5 for each period

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Study Director, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Paris, France

REFERENCES:
- [Result] Hurbin F, Boulenc X, Daskalakis N, Farenc C, Taylor T, Bonneau D, Lacreta F, Cheng S, Sultan E. Clopidogrel pharmacodynamics and pharmacokinetics in the fed and fasted state: a randomized crossover study of healthy men. J Clin Pharmacol. 2012 Oct;52(10):1506-15. doi: 10.1177/0091270011419852. Epub 2011 Nov 29. PMID 22128201